CLINICAL TRIAL: NCT03108079
Title: Bladder Morphology Using 2 Different Catheter Designs Foley Catheter vs. Cystosure Urinary Access System
Brief Title: Bladder Morphology Using 2 Different Catheter Designs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Pelvic Floor Institute (Other)
Collaborators: Cystosure (Unknown); Innovative Research Inc. (Unknown)
Responsible Party: Principal Investigator, Lennox Hoyte, MD, Principal Investigator, The Pelvic Floor Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 03082017
Record Dates: First submitted 2017-03-30; First posted 2017-04-11 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Urologic Injuries; Urologic Diseases; Bladder Infection; Urinary Tract Infections; Mucosal Inflammation; Mucosal Infection; Bladder Injury; Catheter-Related Infections; Catheter Complications; Catheter; Infection (Indwelling Catheter); Pelvic Floor Disorders; Urinary Incontinence
Keywords: Urologic Injuries; Urologic Diseases; Bladder Infection; Urinary Tract Infections; Mucosal Inflammation; Mucosal Infection; Bladder Injury; Catheter Related Infections; Catheter Complications; Catheter Infection; Indwelling Catheter; Pelvic Floor Disorders; Urinary Incontinence
MeSH Terms: conditions — Urologic Diseases; Cystitis; Urinary Tract Infections; Mucositis; Catheter-Related Infections; Infections; Pelvic Floor Disorders; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Female patients seen at the Pelvic Floor Institute will be offered participation in the study. The study will consist of a pelvic floor MRI at no cost to them or their payors. Women who agree to participate will undergo a standard high resolution, thin slice pelvic floor static/dynamic MRI study, first with a full bladder, and after the bladder is emptied. Bladder filling and drainage will be performed sequentially, using each of the 2 catheter types (A and B above) in sequence. During bladder emptying, a cine video scan will be taken at the midsagittal plane to show the dynamics of the bladder fluid and walls during emptying. Each subject will serve as their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Arm 1 (Other): Women who agree to participate will undergo a standard high resolution, thin slice pelvic floor static/dynamic MRI study, first with a full bladder, and after the bladder is emptied. Bladder filling and drainage will be performed sequentially, using each of the 2 catheter types (Cystosure Urinary Access Catheter and Foley Catheter). During bladder emptying, a cine video scan will be taken at the midsagittal plane to show the dynamics of the bladder fluid and walls during emptying. Each subject will serve as their own control.
  Interventions are listed in the "Interventions" Section.
  Interventions: Device: Cystosure Urinary Access System; Device: Foley Catheter

INTERVENTIONS:
Device: Cystosure Urinary Access System — 1. Demonstrate the 3D bladder wall anatomy with 300 cc of fluid infused with each of the following bladder drainage mechanisms
     1. The traditional Foley catheter (Catheter A)
     2. The novel FDA approved Cystosure catheter (Catheter B)
  2. Compare the fluid flow pattern during bladder drainage for
     1. The traditional Foley catheter (Catheter A)
     2. The novel FDA approved Cystosure catheter (Catheter B)
  3. Compare the 3D bladder wall anatomy after emptying the bladder with
     1. The traditional Foley catheter (Catheter A)
     2. The novel FDA approved Cystosure catheter (Catheter B)
  Other Names: Emmy Medical Cystosure Urinary Access System 10-200
Device: Foley Catheter — 1. Demonstrate the 3D bladder wall anatomy with 300 cc of fluid infused with each of the following bladder drainage mechanisms
     1. The traditional Foley catheter (Catheter A)
     2. The novel FDA approved Cystosure catheter (Catheter B)
  2. Compare the fluid flow pattern during bladder drainage for
     1. The traditional Foley catheter (Catheter A)
     2. The novel FDA approved Cystosure catheter (Catheter B)
  3. Compare the 3D bladder wall anatomy after emptying the bladder with
     1. The traditional Foley catheter (Catheter A)
     2. The novel FDA approved Cystosure catheter (Catheter B)
  Other Names: BARD Medical Foley Catheter

SUMMARY:
Demonstrate and compare the 3D morphology of the bladder wall in full and drained states with 2 different kinds of bladder catheters in place. (Foley Catheter vs. Cystosure Catheter)

DETAILED DESCRIPTION:
The Foley catheter has been the mainstay of bladder drainage for many decades. There has been little design change despite risks associated with Foley catheter use including cather associated Urinary Tract Infections(UTIs). However, recent incentives and penalties related to iatrogenic bladder infections have encouraged healthcare providers to search for ways to decrease catheter-associated infections. Data suggests that the design of the traditional Foley catheter may be responsible for bladder mucosal injury due to contact with the drainage tip, which in turn contribute to bladder infections associated with long term indwelling Foley catheter usage. The Cystosure catheter is an FDA approved bladder drainage device, with a shortened drainage port, designed to avoid contact with the bladder mucosa. It is postulated that the lack of contact with the mucosa would decrease mucosal injury, possibly leading to decreased incidence of catheter related bladder infections. Early sheep bladder microscopy studies have suggested that the Cystosure catheter produces significantly less mucosal injury compared to the Foley catheter following a short period of indwelling bladder catheterization. The present study is designed to compare bladder wall geometry around the drainage balloon in the Foley versus the Cystosure drainage catheters in living women. It is hypothesized that the "tip-less" cystosure catheter will have a smoother, more continuous bladder contour around the drainage port, compared to the traditional Foley catheter tip.

ELIGIBILITY:
Inclusion Criteria:

* Pelvic Floor Institute patients aged between 21 and 70 years of age, who are able to speak and understand English, who are not currently pregnant, or had a pregnancy in the previous 6 months.

Exclusion Criteria:

* Women with claustrophobia or any contraindication to undergoing an MRI scan will be excluded. Similarly, women with hip, knee, or shoulder replacements will be excluded because of the need for urethral catheterization. Women with significant mitral valve prolapse will also be excluded for the same reason. Women with history of 3 or more culture-documented UTIs over the last 12 months will be excluded. Women who are unable or unwilling to give informed consent will also be excluded. Women who are unable to tolerate 300 cc of fluid in the bladder will be excluded. Women with a nitrite-positive urinalysis at the time of study enrollment will be excluded until they can demonstrate a negative urine culture.

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients in the trial must be female.
Enrollment: 3 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2017-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Bladder shape after emptying | 1 month
  Bladder shape after emptying using both catheters will be assessed. The 3D reconstructed images will be compared to determine if there are any differences in bladder shape in full and empty states between the 2 catheter types.

CONTACTS AND LOCATIONS:
Overall Officials: Lennox Hoyte, MD, MSEECS, Principal Investigator — The Pelvic Floor Institute
Locations (1):
- The Pelvic Floor Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No